CLINICAL TRIAL: NCT05069857
Title: Neoadjuvant Personalized Anti-PD-1 Therapy With Combination of Anti-VEGFR Therapy in Locally Advanced and Resectable Oral Squamous Cell Carcinoma: A Randomized Controlled Phase II Trial
Brief Title: Neoadjuvant Personalized Anti-PD-1 and Anti-VEGFR Therapy in OSCC Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Lai-ping Zhong, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Icemelting-2
Record Dates: First submitted 2021-09-24; First posted 2021-10-06 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Oral Squamous Cell Carcinoma; Neoadjvant Therapy; Anti-PD-1; Anti-VEGFR
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant arm (Experimental): The patients received three cycles of neoadjuvant therapy, with 14 days each. Dosage and administration: 200mg Carrelizumab intravenously on the first day of each cycle; Apatinib orally 250mg once a day from the first day of each cycle until the 9th day of the third cycle. Then the patients received the standard treatment of surgery and postoperative adjuvant therapy of radiotherapy or chemoradiotherapy.
  Interventions: Drug: Camrelizumab (anti-PD-1 inhibitor); Drug: Apatinib (anti-VEGFR inhibitor)
- Control arm (No Intervention): The patients received the standard treatment of surgery and postoperative adjuvant therapy of radiotherapy or chemoradiotherapy.

INTERVENTIONS:
Drug: Camrelizumab (anti-PD-1 inhibitor) — The patients will receive three cycles of Camrelizumab, with 14 days each. 200mg of Carrelizumab will be used intravenously on the first day of each cycle.
  Arms: Neoadjuvant arm
Drug: Apatinib (anti-VEGFR inhibitor) — The patients will receive Apatinib orally 250mg once a day from the first day of each cycle until the 9th day of the third cycle.
  Arms: Neoadjuvant arm

SUMMARY:
To evaluate the efficacy of neoadjuvant anti-PD-1 plus anti-VEGFR therapy for patients with locally advanced and resectable oral squamous cell carcinoma, and the CPS>10 in the biopsy samples.

DETAILED DESCRIPTION:
In the previous "Icemelting" trial, neoadjuvant anti-PD-1 plus anti-VEGFR therapy was used in 20 patients with locally advanced and resectable oral squamous cell carcinoma (OSCC), and the neoadjuvant therapy was well-tolerated, with no grade 3-4 toxicity. The MPR rate was 40% (8/20), including 5% (1/20) pathological complete response; furthermore, in the patients with CPS>10, the MPR rate was 100%. As we know, the MPR might transfer to survival benefit in the patients received neoadjuvant therapy. Therefore, in this randomized phase II trial, we aimed to evaluate the survival benefit of neoadjuvant anti-PD-1 plus anti-VEGFR therapy in the patients with locally advanced OSCC and CPS>10 (Icemelting-2 trial). A total of 46 patients will be enrolled in this trial, and the primary endpoint is 2-year disease-free survival rate. The neoadjuvant therapy arm will receive three cycles of Carrelizumab plus Apatinib with 14 days each, followed by the standard treatment of surgery and postoperative adjuvant therapy. The control arm will received the standard treatment of surgery and postoperative adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 75
2. Gender: Male and female
3. ECOG Score: 0-2
4. Histologically confirmed primary oral squamous cell carcinoma (including tongue, gingival, buccal, oral base, hard palate, posterior molar area)
5. Clinical stage III/IVA (cT1-2/N1-2/M0 or cT3-4a/N0-2 /M0, AJCC 8th)
6. The combined positive score (CPS score) of PD-L1 expression > 10
7. Has signed informed consent

Exclusion Criteria:

1. Toxicity of ≥ grade 2 (CTCAE 5.0) that has not subsided due to previous anticancer therapy
2. Obvious cardiovascular abnormalities (such as myocardial infarction, superior vena cava syndrome, ≥ grade 2 heart disease diagnosed according to the NYHA classification criteria within 3 months prior to enrollment)
3. Active severe clinical infection (> NCI-CTCAE Version 5.0 level 2 infection)
4. Uncontrollable hypertension (systolic blood pressure > after antihypertensive medication; 150mmHg and/or diastolic blood pressure > 90mmHg) or clinically significant (such as activity) cardiovascular disease, such as cerebrovascular accident (≤ 6 months before screening), myocardial infarction (≤ 6 months before screening), unstable angina, congestive heart failure rated class II or above by NYHA, or severe arrhythmias that cannot be controlled or have a potential impact on trial treatment
5. Blood routine examination: WBC < 3,000/mm3, hemoglobin < 8g/L, platelet < 80,000/mm3
6. Liver function: ALAT/ASAT > 2.5 times the normal upper limit, bilirubin > 1.5 times the normal upper limit
7. Renal function: serum creatinine > 1.5 times the normal upper limit
8. Has a history of maxillofacial and neck radiotherapy
9. Pregnant or lactating women
10. Participation in other clinical studies within 30 days prior to enrollment
11. Other conditions that the investigator considers inappropriate for participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
2-year disease-free survival rate | 24 months
  Disease-free survival was calculated from the date of randomization to tumor recurrence or death from any cause.

SECONDARY OUTCOMES:
2-year overall survival rate | 24 months
  Overall survival was calculated from the date of randomization to death from any cause.
Major pathological response | 3 months
  The major pathological response (MPR): the percentage of tumor cells before and after treatment was compared according to biopsy specimens before neoadjuvant therapy and pathological specimens after surgery; the percentage of residual viable tumor (RVT) cells was evaluated on resected tumor slides. MPR was defined as ≤ 10% RVT%.

CONTACTS AND LOCATIONS:
Overall Officials: Lai-ping Zhong, MD, PhD, Principal Investigator — Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The study protocol and the primary study report might be shared depending on the condition of trial completion.